CLINICAL TRIAL: NCT06373068
Title: A Retrospective Study of the Association of Different Levels of Resuscitation Orders and Mortality in ICU Patients.
Brief Title: Association Between Resuscitation Orders and Mortality in ICU Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sandra Jonmarker, Consultant in Anaesthesia and Intensive care, Ph D, Karolinska Institutet
Other Study IDs: Resuscitation Orders ICU
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness
Keywords: Resuscitation orders
MeSH Terms: conditions — Critical Illness | interventions — Resuscitation Orders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Full code: Patients without any restrictions on the types of treatments available, such as cardiopulmonary resuscitation, intubation, various life support measures, surgery, etc., if indicated.
  Interventions: Other: Resuscitation orders
- Simple Do-Not-Attempt-Resuscitation: The only treatment limitation in patient care is cardiopulmonary resuscitation in case of a cardiac arrest. All other indicated devices or treatments may still be utilized.
  Interventions: Other: Resuscitation orders
- Do not attempt resuscitation with limited scope: The treatment limitation in patient care includes not performing cardiopulmonary resuscitation and also involve additional limitations, typically including various life support measures.
  Interventions: Other: Resuscitation orders

INTERVENTIONS:
Other: Resuscitation orders — Resuscitation orders, commonly referred to as Code Status, communicate to the healthcare team the specific medical interventions that patients will receive while hospitalised. These orders are issued by a doctor and require confirmation by at least one other licensed medical professional

SUMMARY:
The hypothesis of the study is that a resuscitation order other than full code is associated with increased mortality among critically ill patients. By incorporating conventional variables associated with death such as age, sex, and Simplified Acute Physiological Score, as well as including the new Clinical Frailty Scale in a statistical model, the aim is to investigate whether there is still an increased risk of death that remains unexplained.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU

Exclusion Criteria:

* Second or subsequent admission to ICU during the study period.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients admitted to the intensive care unit during 2023 and 2024
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 365 days
  Hazard ratio of death

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jonmarker, Principal Investigator — Stockholm South General Hospital
Locations (1):
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The privacy of the data is protected under Swedish law, and the original patient data will be stored in a de-identified form for 10 years in accordance with Karolinska Institute regulations. Use of the de-identified data for research purposes beyond those specified in this registration may be considered, but requires additional approval from the Swedish Ethics Committee.